CLINICAL TRIAL: NCT04717427
Title: Integrated Longitudinal Studies to Identify Biomarkers and Therapeutic Strategies for Sturge-Weber Syndrome
Brief Title: Longitudinal Studies to Identify Biomarkers for Sturge-Weber Syndrome
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of California, San Francisco (Other); Wayne State University (Other); Duke University (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Children's Hospital Medical Center, Cincinnati (Other); Boston Children's Hospital (Other); Nationwide Children's Hospital (Other); Sturge-Weber Foundation (Other)
Responsible Party: Principal Investigator, Jeffrey A Loeb, Professor, University of Illinois at Chicago
Other Study IDs: 2020-1165
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Sturge-Weber Syndrome
MeSH Terms: conditions — Sturge-Weber Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individuals with Sturge-Weber Syndrome (SWS) sometimes have brain involvement which can result in seizures, stroke-like episodes and neurologic deficits. The purpose of this study is to integrate longitudinal clinical data, radiological data, and blood biomarkers of Sturge-Weber syndrome patients.

The research aims are:

1. To integrate longitudinal clinical data, radiological data, and blood biomarkers of Sturge-Weber syndrome patients.
2. Identify plasma and imaging biomarkers sensitive to exacerbation of clinical symptoms including seizures, headaches, or stroke-like episodes.
3. For enrolled patients who present with severe neurological symptoms screen blood samples for inflammatory changes.

The target enrollment for this study is about 250 individuals diagnosed with Sturge-Weber Syndrome. The goal of this study is to understand more about Sturge-Weber Syndrome, the possible treatments for this disease, and identify targets for clinical trials. Those participating in the database will be asked to consent to blood draws.

DETAILED DESCRIPTION:
Aim 1: Develop a longitudinal database of patients with SWS Clinical sites will collect longitudinal data retrospectively on measures of clinical symptoms and medications/treatments for study subjects who participated in the existing BVMC2/SWF registry and consent to participate in BVMC3 study. Retrospective data will be used to create a longitudinal dashboard where practitioners can identify predictors of atrisk patients who are most likely to have a serious neurological symptom and the current treatments. Prospective data collection: Clinical sites will collect longitudinal data prospectively for at-risk patients who present with a new, severe neurological symptom.

Aim 2: Examine longitudinal Quantitative MRI Baseline MRI datasets will be collected and Limited Data Sets (LDS) will be generated and uploaded to a central imaging database from all participating centers. Subsequent MRI scans will be collected for patients who experience acute exacerbation of clinical symptoms, including seizures, headaches, or stroke-like episodes. Integrated imaging data, detailed treatment data, and detailed clinical data including neurological symptoms, seizures, and headache history will be analyzed.

Aim 3: Collect and Store Blood Samples for Analysis All patients enrolled in BVMC3 study will have blood samples sent to and stored at University of California San Francisco (UCSF). Enrolled patients presenting with stroke-like episodes, stroke, headache, or seizure will have a second blood sample taken at the time of the neurologic symptom and a third sample taken 6 months later, or even later if symptoms have not resolved within 6 months. Multiplex angioma and inflammatory marker array will be assessed on all 3 samples from patients at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MRI-documented unilateral or bilateral leptomeningeal angiomas with or without neurological symptoms including seizures, headaches, and stroke-like episodes
* Patients of any age
* Availability of longitudinal clinical and imaging data from all patient EHR records
* Consent to being followed prospectively throughout the course of the study
* Willing to provide blood samples
* Inclusion criteria to trigger entry into Aim 1B: severe seizures, headaches, or stroke-like episodes

Exclusion Criteria:

* Persons without physician diagnosed SWS
* Persons unwilling to sign informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Assemble a cohort of 250 patients with standardized phenotyping/diagnosis to collect standardized longitudinal clinical and radiological data and obtain blood samples at enrollment. We anticipate 25% of 250 enrolled patients will have serious neurological symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Natural history of disease progression. | 4 years
  Integrative aspect that examines longitudinal associations of clinical symptoms, radiological disease progression, medical treatments, and blood biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Loeb, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - University of Illinois At Chicago, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio